CLINICAL TRIAL: NCT05660473
Title: Pediatric-inspired Regimen Combined With Venetoclax for Adolescent and Adult Patients With de Novo Philadelphia Chromosome-Negative Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022052
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: Philadelphia Chromosome-Negative; Acute Lymphoblastic Leukemia; Adolescent and Adult; Pediatric-inspired Regimen; Venetoclax
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Daunorubicin; Cyclophosphamide; pegaspargase; Prednisone; Cytarabine; Mercaptopurine; Dexamethasone; Methotrexate; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pediatric-inspired Regimen Combined With Venetoclax (Experimental): Induction therapy is administered as follows：Vincristine (VCR) 1.4 mg/m2 (maximum dose 2 mg) IV on D1,8,1,5,22; Daunorubicin (DNR) 30 mg/m2/day IV on D1-3; Cyclophosphamide (CTX) 1200 mg/m2 IV on D1,15; Pegaspargase 2500u/m2 IM on D5; Prednisone 1 mg/kg/d PO on D1-14, 0.5 mg/kg/d PO on D15-28; Venetoclax 100 mg PO on D6，200 mg on D7, 400mg on D8-14, All patients underwent bone marrow aspiration on day 14 during induction. Patients with bone marrow blasts ≥10% on day 14 of induction received 7 additional days of Venetoclax on day 15-22. Consolidation therapy is a combination of multi-drug pediatric-inspired regimen chemotherapy and Venetoclax. Maintenance therapy consisted of a monthly VMMP regimen (vincristine, mercaptopurine, methotrexate, prednisone) continuing until 3 years for male and 2.5 years for female patients.
  Interventions: Drug: Vincristine; Drug: Daunorubicin; Drug: Cyclophosphamide; Drug: Pegaspargase; Drug: Prednisone; Drug: Cytarabine; Drug: 6-mercaptopurine; Drug: Dexamethasone; Drug: Methotrexate; Drug: Venetoclax

INTERVENTIONS:
Drug: Vincristine — Anti-tumor alkaloids
Drug: Daunorubicin — Anthracycline
Drug: Cyclophosphamide — Alkylating agent
Drug: Pegaspargase — Polyethylene glycol (PEG) conjugated to L-asparaginase
Drug: Prednisone — Glucocorticoids
Drug: Cytarabine — Pyrimidine antimetabolites
Drug: 6-mercaptopurine — Cell cycle-specific antitumor drug
Drug: Dexamethasone — Glucocorticoids
Drug: Methotrexate — Antifolate antineoplastic drug
Drug: Venetoclax — Selective inhibitor of B-cell lymphoma 2 (Bcl-2)

SUMMARY:
The pediatric-inspired regimen has greatly improved the prognosis of adult patients with with Philadelphia chromosome-negative acute lymphoblastic leukemia (Ph- ALL), but relapse remains a great challenge. Venetoclax (Ven) is an oral, selective inhibitor of B-cell lymphoma 2 (Bcl-2). Although this drug is currently used primarily for acute myeloid leukemia, in vitro as well as small cohort studies suggest a effect in acute lymphoblastic leukemia. This study proposes to combine pediatric-inspired regimen with venetoclax for the treatment of adult patients with Ph- ALL, aiming to improve the MRD-negative complete remission rate measured by flow cytometry after induction and to reduce relapse, thus further improving patients overall survival.

ELIGIBILITY:
Inclusion Criteria:

* De novo and primary Ph/BCR-ABL1 negative acute lymphoblastic leukemia diagnosed by the bone marrow cytomorphology, immunophenotyping, cytogenetics and molecular biology according to WHO classification
* Age: 14 -60 years
* Male or female
* ECOG Performance Status 0-2
* Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤5 x ULN if leukemic involvement of the liver is present; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; normal electrolytes: Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN; Cardiac color Doppler ultrasound ejection fraction ≥ 45%;
* Subject has provided written informed consent prior to any screening procedure

Exclusion Criteria:

* Burkitt lymphoma/leukemia
* Acute Leukemia of Ambiguous Lineage
* Female patients who are pregnant or breast feeding
* Uncontrolled active serious infections that could, in the investigator's opinion, potentially interfere with the completion of treatment
* History of pancreatitis
* Poorly controlled diabetes, defined as glycosylated hemoglobin (HbA1c) values of >7.5%. Patients with preexisting, well-controlled diabetes are not excluded
* History of active gastrointestinal bleeding within the last 6 months
* History of arterial/venous thrombosis within the last 6 months
* Known HIV seropositivity
* Any serious psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
MRD-negative complete remission rate measured by flow cytometry | After induction (4 week)

SECONDARY OUTCOMES:
Complete remission (CR) rate | After 2 cycles of chemotherapy, an expected average of 3 months
Overall survival (OS) | Up to 5 years post-registration
  From the date of registration to the date of death resulting from any cause
Relapse free survival (RFS) | Up to 5 years post-registration
  From the date of complete remission(CR) until the date of documented relapse or death due to any cause or the last follow-up day
Disease-free Survival (DFS) | Up to 5 years post-registration
  From CR1 to relapse, death from any cause or last follow-up
The rate of adverse events | An expected average of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No